CLINICAL TRIAL: NCT01890967
Title: A Phase 2 Efficacy and Safety Dose-Ranging Study of LY3015014 in Patients With Primary Hypercholesterolemia
Brief Title: A Study of LY3015014 in Participants With High Cholesterol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14853; I5S-MC-EFJE (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Hypercholesterolemia
Keywords: low density lipoprotein, heterozygous familial hypercholesterolemia, polygenic hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — frovocimab; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Simvastatin; Rosuvastatin Calcium; Pravastatin; Lovastatin; Fluvastatin; pitavastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 20 mg LY3015014 Q4W (Experimental): 20 milligrams (mg) LY3015014 given subcutaneously (SC) once every 4 weeks (Q4W) for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
  Interventions: Drug: LY3015014; Drug: Statin; Drug: Ezetimibe
- 120 mg LY3015014 Q4W (Experimental): 120 mg LY3015014 given SC Q4W for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
  Interventions: Drug: LY3015014; Drug: Statin; Drug: Ezetimibe
- 300 mg LY3015014 Q4W (Experimental): 300 mg LY3015014 given SC Q4W for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
  Interventions: Drug: LY3015014; Drug: Statin; Drug: Ezetimibe
- 100 mg LY3015014 Q8W (Experimental): 100 mg LY3015014 given SC once every 8 weeks (Q8W) for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
  Interventions: Drug: LY3015014; Drug: Statin; Drug: Ezetimibe
- 300 mg LY3015014 Q8W (Experimental): 300 mg LY3015014 given SC Q8W for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
  Interventions: Drug: LY3015014; Drug: Statin; Drug: Ezetimibe
- Placebo Q4W (Placebo Comparator): Placebo given SC Q4W for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
  Interventions: Drug: Placebo; Drug: Statin; Drug: Ezetimibe

INTERVENTIONS:
Drug: LY3015014 — Administered SC
  Arms: 100 mg LY3015014 Q8W; 120 mg LY3015014 Q4W; 20 mg LY3015014 Q4W; 300 mg LY3015014 Q4W; 300 mg LY3015014 Q8W
Drug: Placebo — Administered SC
  Arms: Placebo Q4W
Drug: Statin — Administered orally
  Other Names: atorvastatin; simvastatin; rosuvastatin; pravastatin; lovastatin; fluvastatin; pitavastatin
Drug: Ezetimibe — Administered orally

SUMMARY:
This study is designed to define the amount and duration of cholesterol lowering and to assess the safety and tolerability of different dose regimens of LY3015014 in participants with high cholesterol. The study will also investigate how the body processes the drug and how the drug affects the body. Participants will remain on a stable diet and will continue taking cholesterol-lowering medications (statins with or without ezetimibe). After signing the informed consent document, the participant will complete a screening/run-in period that will last at most 8 weeks. Then, the treatment period will last approximately 16 weeks. After the treatment period, the participants will complete a follow-up period lasting approximately 8 weeks for a total study duration ranging from approximately 25 to 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with high low density lipoprotein (LDL) cholesterol
* Are on stable daily dose of a statin or have a history of statin intolerance
* Men with a partner who can become pregnant must agree to use barrier protection during sexual intercourse to prevent pregnancies
* Women who cannot become pregnant, or women who are not pregnant or breast feeding and agree to use a reliable method of birth control to prevent pregnancies

Exclusion Criteria:

* Have high cholesterol due to another disease or have a rare and serious form of hereditary high cholesterol
* Have had recent heart attack, stroke, blood clot or heart surgery, have planned heart or blood vessel surgery, or has a heart that does not pump sufficiently well
* Have poorly controlled high blood pressure
* Have diabetes that requires an injectable medication (including insulin), or have diabetes that is poorly controlled
* Have thyroid blood test that is outside normal range
* Have a history of adrenal gland disorder
* Have a history of vitamin E deficiency or fat malabsorption syndrome
* Have poor kidney function
* Have active liver or gall bladder disease, history of hepatitis or liver blood tests that are high
* Have a history of muscle disease including muscle damage from a medicine or muscle blood test that is high
* Are anemic (low red blood cell counts)
* Have a history of allergy or intolerance to other antibody medications
* Have a history of human immunodeficiency virus infection (HIV) infection
* Are likely to have a major operation or be hospitalized during the study
* Have chronic alcohol or drug abuse or dependency
* Have or suspected to have any cancer or malignant tumor
* Have an active serious infection
* Have started or stopped taking a statin or ezetimibe medication, or changed statin dose regimen recently
* Are on a statin regimen other than daily dosing (for example, an every-other-day statin regimen)
* Have recently used simvastatin (highest dose level), fibrates, bile acid binders, niacin, probucol, or over-the-counter/health food preparations to lower cholesterol (such as red yeast rice, fish oil, omega 3 fatty acid)
* Have undergone LDL apheresis in the past 1 year
* Have recently used steroids, cyclosporine or isotretinoin
* Have recently used an immunosuppressive therapy
* Have recently received treatment with another antibody medication
* Are currently using medications injected into the skin , except for single injections (for example flu vaccines) or injections into muscles
* Are currently on a prescription or over-the-counter medicine for weight loss or are on a very low carbohydrate diet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Encino, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Safety Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bossier City, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
- Canada (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kamloops, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brampton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gatineau, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Marc-des-Carrieres, Quebec
- Czechia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Český Krumlov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hodonín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Svitavy
- Denmark (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalborg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esbjerg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hellerup
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hvidovre
- Japan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Netherlands (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Groningen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maastricht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Utrecht
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Q4W: Placebo given subcutaneously (SC) once every 4 weeks (Q4W) for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
- 20 mg LY3015014 Q4W: 20 milligrams (mg) LY3015014 given SC Q4W for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
Period: Overall Study
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Started | 88 | 88 | 88 | 88 | 87 | 88
Received at Least One Dose of Study Drug | 87 | 87 | 86 | 86 | 86 | 87
Completed | 78 | 77 | 78 | 77 | 77 | 75
Not Completed | 10 | 11 | 10 | 11 | 10 | 13
Not completed — Adverse Event | 3 | 3 | 3 | 2 | 1 | 7
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 3 | 3 | 2 | 4 | 1
Not completed — Sponsor Decision | 2 | 0 | 1 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 3 | 4 | 2 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- 20 mg LY3015014 Q4W: 20 mg LY3015014 given subcutaneously SC Q4W for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
- 100 mg LY3015014 Q8W: 100 mg LY3015014 given SC Q8W for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
- Total: Total of all reporting groups
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W | Total
Number analyzed (Participants) | 87 | 87 | 86 | 86 | 86 | 87 | 519
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (11.2) | 57.2 (9.4) | 57.1 (12.4) | 59.7 (9.4) | 59.6 (8.1) | 58.7 (10.1) | 58.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 41 | 39 | 36 | 43 | 241
  Male | 47 | 45 | 45 | 47 | 50 | 44 | 278
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 3 | 1 | 2 | 13
  Not Hispanic or Latino | 56 | 53 | 52 | 51 | 51 | 52 | 315
  Unknown or Not Reported | 28 | 32 | 32 | 32 | 34 | 33 | 191
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 25 | 22 | 21 | 25 | 21 | 23 | 137
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 6 | 1 | 6 | 5 | 23
  White | 60 | 61 | 59 | 60 | 58 | 58 | 356
  More than one race | 1 | 0 | 0 | 0 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Canada | 13 | 17 | 13 | 15 | 17 | 19 | 94
  Netherlands | 16 | 16 | 17 | 11 | 13 | 15 | 88
  Czech Republic | 5 | 2 | 3 | 4 | 5 | 4 | 23
  Puerto Rico | 2 | 0 | 1 | 1 | 0 | 1 | 5
  United States | 25 | 23 | 26 | 26 | 22 | 21 | 143
  Japan | 17 | 18 | 18 | 17 | 18 | 18 | 106
  Denmark | 3 | 4 | 5 | 6 | 6 | 5 | 29
  Poland | 6 | 7 | 3 | 6 | 5 | 4 | 31
Serum LDL Cholesterol Beta Quantification [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 136.5 (39.6) | 134.1 (42.4) | 134.0 (40.7) | 132.1 (42.3) | 135.2 (41.2) | 146.0 (60.5) | 136.3 (45.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C)
Description: Least square (LS) Means was calculated using analysis of covariance (ANCOVA) adjusted for disease classification, statin dose, baseline LDL-C measurement. Percent change from baseline response is the dependent variable.
Time Frame: Baseline, Week 16
Population: Modified Intent to Treat (mITT) is defined as all patients in the ITT population who had at least one baseline measurement and one post-randomization measurement of the variable that is analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Groups:
- 20 mg LY3015014 Q4W: 20 mg LY3015014 given SC Q4W for 16 weeks.
  Participants will remain on stable diet and physician-prescribed statin therapy, if tolerated, with or without ezetimibe.
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Number analyzed (Participants) | 79 | 75 | 78 | 76 | 73 | 73
Percentage change | 7.6 (2.27) | -14.9 (2.39) | -40.5 (2.31) | -50.5 (2.30) | -14.9 (2.35) | -37.1 (2.44)

2. Secondary Outcome: Percentage Change From Baseline in LDL-C, Total Cholesterol (TC), High-Density Lipoprotein Cholesterol (HDL-C), Triglycerides (TG), Non-HDL-C
Description: LS Mean was calculated using mixed model repeated measures (MMRM) analysis with baseline measurement, disease classification, statin dose, treatment, visit, and treatment by visit interaction included in the model. Percent change from baseline response is the dependent variable.
Time Frame: Baseline, Week 16
Population: mITT is defined as all patients in the ITT population who had at least one baseline measurement and one post-randomization measurement of the variable that is analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Number analyzed (Participants) | 86 | 86 | 86 | 85 | 86 | 87
Percentage change
  LDL-C: number analyzed (Participants) | 78 | 77 | 78 | 78 | 77 | 73
  LDL-C | 5.9 (2.13) | -18.0 (2.18) | -46.4 (2.15) | -56.5 (2.14) | -18.4 (2.14) | -42.2 (2.21)
  TG: number analyzed (Participants) | 78 | 78 | 80 | 79 | 76 | 74
  TG | 3.5 (3.26) | -6.1 (3.35) | -7.2 (3.25) | -15.1 (3.26) | -7.2 (3.29) | -10.6 (3.35)
  TC: number analyzed (Participants) | 78 | 78 | 80 | 79 | 76 | 74
  TC | 3.5 (1.44) | -10.5 (1.47) | -27.8 (1.44) | -34.1 (1.44) | -11.0 (1.45) | -24.6 (1.48)
  HDL-C: number analyzed (Participants) | 78 | 78 | 80 | 79 | 76 | 74
  HDL-C | 1.6 (1.58) | 4.5 (1.60) | 7.3 (1.57) | 8.8 (1.58) | 4.5 (1.59) | 8.4 (1.61)
  Non-HDL-C: number analyzed (Participants) | 78 | 78 | 80 | 79 | 76 | 74
  Non-HDL-C | 4.9 (1.83) | -16.1 (1.86) | -39.3 (1.83) | -48.9 (1.83) | -16.1 (1.84) | -35.8 (1.88)

3. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein A1 (Apo A1), Apolipoprotein B (Apo B)
Description: LS Mean was calculated using MMRM analysis with baseline measurement, disease classification, statin dose, treatment, visit, and treatment by visit interaction included in the model. Percent change from baseline response is the dependent variable.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Number analyzed (Participants) | 86 | 84 | 84 | 85 | 85 | 87
Percentage change
  Apo A1: number analyzed (Participants) | 78 | 77 | 78 | 78 | 75 | 73
  Apo A1 | 0.3 (1.40) | 2.4 (1.43) | 6.5 (1.41) | 6.2 (1.41) | 3.8 (1.43) | 5.8 (1.44)
  Apo B: number analyzed (Participants) | 78 | 77 | 78 | 78 | 75 | 73
  Apo B | 4.2 (2.23) | -16.6 (2.32) | -34.9 (2.28) | -46.8 (2.25) | -16.0 (2.25) | -31.9 (2.31)

4. Secondary Outcome: Percentage Change From Baseline in Lipoprotein(a) [Lp(a)]
Description: Data was log-transformed for MMRM analysis, with change from baseline as the dependent variable, and baseline measurement, disease classification, statin dose, treatment, visit, and treatment by visit interaction included as independent variables. Percentage change from baseline in the original scale was then back-calculated from the log-transformed MMRM analysis.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Number analyzed (Participants) | 68 | 71 | 73 | 75 | 70 | 68
Percentage Change | -0.31 (0.0436) | -16.63 (0.0442) | -19.02 (0.0427) | -37.29 (0.0420) | -7.54 (0.0427) | -21.01 (0.0437)

5. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (hsCRP)
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Number analyzed (Participants) | 78 | 75 | 80 | 78 | 76 | 73
Percentage change | 0.5 (0.70) | -0.2 (0.72) | 1.6 (0.69) | -0.3 (0.70) | -0.3 (0.70) | -0.7 (0.72)

6. Secondary Outcome: Number of Participants Who Develop Treatment Emergent Anti-LY3015014 Antibodies
Time Frame: Baseline through Week 24
Population: All randomized participants who received at least one dose of study treatment and had evaluable data.
Measure: Number; unit: Participants
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Number analyzed (Participants) | 86 | 86 | 86 | 85 | 86 | 87
Participants | 4 | 6 | 10 | 5 | 4 | 3

7. Secondary Outcome: Percentage Change From Baseline in Total Proprotein Convertase Subtilisin/Kexin Type 9 Antibody (PCSK9) Levels
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Number analyzed (Participants) | 77 | 76 | 79 | 79 | 75 | 75
Percentage change | 14.6 (13.66) | 9.1 (14.00) | 86.4 (13.65) | 130.6 (13.63) | 21.8 (13.63) | 41.0 (13.63)

8. Secondary Outcome: Percentage Change From Baseline in Free Proprotein Convertase Subtilisin/Kexin Type 9 Antibody (PCSK9) Levels
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Number analyzed (Participants) | 77 | 72 | 76 | 75 | 70 | 72
Percentage change | 9.9 (5.59) | -16.3 (5.81) | -36.6 (5.67) | -68.0 (5.71) | -4.4 (5.80) | -35.2 (5.72)

9. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve at Steady-State (AUC,ss) for LY3015014
Time Frame: Week 12-16 (Q4W) - Predose, Week 8-16 (Q8W) - Predose
Population: All randomly assigned participants who received at least one dose of the study medication and had evaluable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg∙hr/mL
Arm/Group | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Number analyzed (Participants) | 83 | 85 | 82 | 84 | 86
μg∙hr/mL | 1590 (29.2) | 9670 (29.9) | 27300 (26.3) | 7800 (28.5) | 26600 (32.2)

10. Secondary Outcome: Number of Participants With an Injection Site Reaction
Time Frame: Baseline through Week 24
Population: All randomized participants who received at least one dose of study treatment and had evaluable data.
Measure: Number; unit: Participants
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Number analyzed (Participants) | 87 | 87 | 86 | 86 | 86 | 87
Participants | 26 | 42 | 57 | 51 | 36 | 41

ADVERSE EVENTS:
Description: Participants at Risk included all participants who received at least one dose of study drug.
Arm/Group | Placebo Q4W | 20 mg LY3015014 Q4W | 120 mg LY3015014 Q4W | 300 mg LY3015014 Q4W | 100 mg LY3015014 Q8W | 300 mg LY3015014 Q8W
Serious Adverse Events (participants affected / at risk) | 5/87 | 3/87 | 6/86 | 2/86 | 2/86 | 4/87
Other Adverse Events (participants affected / at risk) | 63/87 | 69/87 | 64/86 | 64/86 | 64/86 | 58/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Q4W (N=87) | 20 mg LY3015014 Q4W (N=87) | 120 mg LY3015014 Q4W (N=86) | 300 mg LY3015014 Q4W (N=86) | 100 mg LY3015014 Q8W (N=86) | 300 mg LY3015014 Q8W (N=87)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/47 (0) | 0/45 (0) | 0/45 (0) | 0/47 (0) | 0/50 (0) | 1/44 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/40 (0) | 0/42 (0) | 1/41 (1) | 0/39 (0) | 0/36 (0) | 0/43 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q4W (N=87) | 20 mg LY3015014 Q4W (N=87) | 120 mg LY3015014 Q4W (N=86) | 300 mg LY3015014 Q4W (N=86) | 100 mg LY3015014 Q8W (N=86) | 300 mg LY3015014 Q8W (N=87)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 6 (9) | 6 (6) | 3 (3) | 3 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 6 (6) | 3 (3) | 3 (3) | 1 (1)
Influenza like illness (General disorders) | 6 (8) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Injection site bruising (General disorders) | 4 (4) | 1 (1) | 8 (9) | 2 (2) | 2 (3) | 4 (4)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 9 (10) | 7 (10) | 2 (3) | 3 (3)
Injection site pain (General disorders) | 3 (6) | 15 (20) | 11 (17) | 8 (17) | 7 (13) | 9 (12)
Injection site pruritus (General disorders) | 1 (1) | 4 (6) | 6 (6) | 8 (13) | 2 (2) | 2 (3)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 5 (7) | 6 (10) | 3 (4) | 2 (2)
Bronchitis (Infections and infestations) | 5 (6) | 0 (0) | 2 (2) | 3 (3) | 2 (3) | 3 (3)
Influenza (Infections and infestations) | 3 (3) | 5 (5) | 2 (3) | 3 (3) | 2 (2) | 1 (2)
Nasopharyngitis (Infections and infestations) | 15 (17) | 20 (23) | 22 (22) | 14 (18) | 11 (13) | 15 (18)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (2) | 5 (5) | 7 (8) | 6 (7) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 3 (3) | 6 (6) | 2 (2) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (6) | 9 (10) | 3 (3) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (9) | 6 (8) | 7 (9) | 3 (5) | 6 (6)
Headache (Nervous system disorders) | 6 (7) | 6 (7) | 11 (13) | 8 (11) | 8 (8) | 2 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 5 (6) | 2 (2) | 1 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days